CLINICAL TRIAL: NCT04483531
Title: Odevixibat (A4250) for the Treatment of Progressive Familial Intrahepatic Cholestasis (Expanded Access Program)
Brief Title: Odevixibat for the Treatment of Progressive Familial Intrahepatic Cholestasis
Status: Approved for marketing | Type: Expanded Access
Sponsor: Albireo (Industry)
Responsible Party: Sponsor
Organization: Ipsen (Industry)
Other Study IDs: A4250-014
Record Dates: First submitted 2020-07-13; First posted 2020-07-23 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Progressive Familial Intrahepatic Cholestasis
Keywords: PFIC; pediatric; Cholestasis
MeSH Terms: conditions — Cholestasis, progressive familial intrahepatic 1; Cholestasis | interventions — odevixibat

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: Odevixibat — A4250 is a small molecule and selective inhibitor of IBAT
  Other Names: A4250

SUMMARY:
To provide treatment access to patients with PFIC in the US who have pruritus and elevated serum bile acids and who are not able to enroll in A4250-008 (PEDFIC2) for the following reasons: 1) Do not meet eligibility criteria for PEDFIC 2; 2) Are not able to get to a PEDFIC 2 site for geographical reasons, and 3) Do meet the eligibility criteria for PEDFIC 2 after recruitment has been completed

DETAILED DESCRIPTION:
Eligible patients will be enrolled into this expanded-access program and treated with an oral dose of 120 μg/kg/day of odevixibat and evaluated on an ongoing basis.

ELIGIBILITY:
Inclusion Criteria:

1. A male or female patient of any age, with a clinical diagnosis of PFIC, and with a body weight ≥5 kg at Screening visit
2. Patient must have a clinical diagnosis of PFIC
3. Patient must have clinically confirmed pruritus
4. Patient must have elevated serum bile acid levels, specifically measured to be ≥2 × the upper limit of normal (ULN) prior to start of medication
5. Patient and/or legal guardian must sign informed consent (and assent) as appropriate. Patients who turn 18 years of age (or legal age per country) during

Exclusion Criteria:

1. Patient is expected to have a liver transplant within 6 months of Screening
2. Decompensated liver disease, coagulopathy, history or presence of clinically significant ascites, variceal hemorrhage, and/or encephalopathy
3. International normalized ratio (INR) >1.4 (the patient may be treated with Vitamin K intravenously, and if INR is ≤1.4 at resampling the patient may be started on program medication)
4. Serum ALT >10 × ULN at Screening
5. Serum ALT >15 × ULN at any time point during the last 6 months unless an alternate etiology was confirmed for the elevation
6. Total bilirubin >10 × ULN at Screening
7. Any patient who is pregnant, lactating, or planning to get pregnant
8. Patients who qualify for enrollment in other Phase 2 or Phase 3 trials intended to support marketing approval in PFIC

Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (1):
- Albireo Pharma Inc., Boston, Massachusetts, United States